CLINICAL TRIAL: NCT03937440
Title: The Effect of Deep Neuromuscular Block on the Perioperative Stress Response Reduction and Postoperative Recovery Enhancement in Robot-assisted Stomach Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2019-0205
Record Dates: First submitted 2019-04-28; First posted 2019-05-03 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Stomach Cancer
Keywords: deep neuromuscular block; robot-assisted surgery; stress response; stomach cancer
MeSH Terms: conditions — Stomach Neoplasms; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular block group (Experimental)
  Interventions: Drug: Deep neuromuscular block with 'rocunium®'
- Moderate neuromuscular block group (Experimental)
  Interventions: Drug: Moderate neuromuscular block with 'rocunium®'

INTERVENTIONS:
Drug: Deep neuromuscular block with 'rocunium®' — Rocuronium will be maintained in a arm 1) deep neuromuscular block group or arm 2) moderate neuromuscular block group (control group) according to the assignment. The degree of muscle relaxation is determined by 1 to 2 for post-tetanic count (PTC) in deep neuromuscular group.
  Arms: Deep neuromuscular block group
Drug: Moderate neuromuscular block with 'rocunium®' — Rocuronium will be maintained in a arm 1) deep neuromuscular block group or arm 2) moderate neuromuscular block group (control group) according to the assignment. The degree of muscle relaxation is determined by 1 to 2 for train-of-four (TOF) in moderate neuromuscular group.
  Arms: Moderate neuromuscular block group

SUMMARY:
Stress reactions caused by surgical stimuli can cause sympathetic nervous system activation and increased stress hormones, such as catecholamines, inflammatory cytokines, and pituitary hormones, and insulin resistance. In addition, increased catecholamine levels may exacerbate postoperative outcomes, especially delayed wound recovery, increased cardiovascular and respiratory complications, and immunosuppression. In particular, it is important to reduce the stress response for cancer patients during surgery because they are already immunocompromised status and more vulnerable to perioperative stressful situation. However, there are insufficient results on the benefits of deep neuromuscular block in these patients, although some have reported a reduction of postoperative pain and fewer complications in the deep neuromuscular block compared with moderate neuromuscular block. Therefore, the investigators aim to investigate the difference in the stress response of patients who received conventional moderate neuromuscular block or deep neuromuscular block in robot-assisted gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA Ⅰ - Ⅱ patients between 20 and 65 years undergoing robot-assisted gastric cancer surgery

Exclusion Criteria:

* 1. Patients with neuromuscular disease
* 2. Hypertensive patients with β-blockers
* 3. Diabetic patients receiving insulin therapy
* 4. Patients with severe heart (EF <45%), kidney (GFR <60), liver dysfunction (ALT / AST> 100)
* 5. Patients with obesity (BMI ≥30)
* 6. Do not understand Korean language
* 7. For vulnerable subjects who are unable to obtain consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Difference of stress responses between deep block and moderate block | at baseline (T1)
  Comparison of perioperative stress responses with biomarkers including cortisol, interleukin-6, natural killer cell and HRV between deep neuromuscular block group and moderate neuromuscular group
Difference of stress responses between deep block and moderate block | 90 min after CO2 inflation (T2)
  Comparison of perioperative stress responses with biomarkers including cortisol, interleukin-6, natural killer cell and HRV between deep neuromuscular block group and moderate neuromuscular group
Difference of stress responses between deep block and moderate block | at the end of pneumoperitoneum (about 3 hours after CO2 inflation) (T3)
  Comparison of perioperative stress responses with biomarkers including cortisol, interleukin-6, natural killer cell and HRV between deep neuromuscular block group and moderate neuromuscular group
Difference of stress responses between deep block and moderate block | 1 day after surgery (T4)
  Comparison of perioperative stress responses with biomarkers including cortisol, interleukin-6, natural killer cell and HRV between deep neuromuscular block group and moderate neuromuscular group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea